CLINICAL TRIAL: NCT00493649
Title: Phase II Trial of Adjuvant TC (Docetaxel/Cyclophosphamide) Plus Trastuzumab in HER2-Positive Early Stage Breast Cancer Patients
Brief Title: Adj TC + Herceptin Early Stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-038; 11270 (Other: Sanofi-Aventis)
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TC+H (Experimental): On Day 1 of each 21-day cycle for a total of 4 cycles, patients will receive, in this order: docetaxel (Taxotere) 75 mg/m2 IV (over 1 hour), plus cyclophosphamide (Cytoxan) 600 mg/m2 IV (over 15-30 minutes), plus weekly trastuzumab (Herceptin) 4 mg/kg IV (loading dose, over 90 minutes Day 1, Cycle 1 only) and 2 mg/kg IV (over 30-60 minutes on Days 1, 8, and 15) thereafter.
  Interventions: Drug: Taxotere; Drug: Cytoxan; Drug: Herceptin

INTERVENTIONS:
Drug: Taxotere — On Day 1 of each 21-day cycle for a total of 4 cycles, patients will receive, in this order: docetaxel 75 mg/m2 IV (over 1 hour), plus cyclophosphamide 600 mg/m2 IV (over 15-30 minutes), plus weekly trastuzumab 4 mg/kg IV (loading dose, over 90 minutes Day 1, Cycle 1 only) and 2 mg/kg IV (over 30-60 minutes on Days 1, 8, and 15) thereafter. Once 4 cycles of TC+H have been received, patients will continue with trastuzumab 6 mg/kg every 3 weeks to complete 1 year of anti-HER2 therapy as per the current standard of care. The anticipated time to study completion is 5 years.
  Other Names: docetaxel
Drug: Cytoxan — On Day 1 of each 21-day cycle for a total of 4 cycles, patients will receive, in this order: docetaxel 75 mg/m2 IV (over 1 hour), plus cyclophosphamide 600 mg/m2 IV (over 15-30 minutes), plus weekly trastuzumab 4 mg/kg IV (loading dose, over 90 minutes Day 1, Cycle 1 only) and 2 mg/kg IV (over 30-60 minutes on Days 1, 8, and 15) thereafter. Once 4 cycles of TC+H have been received, patients will continue with trastuzumab 6 mg/kg every 3 weeks to complete 1 year of anti-HER2 therapy as per the current standard of care. The anticipated time to study completion is 5 years.
  Other Names: cyclophosphamide
Drug: Herceptin — On Day 1 of each 21-day cycle for a total of 4 cycles, patients will receive, in this order: docetaxel 75 mg/m2 IV (over 1 hour), plus cyclophosphamide 600 mg/m2 IV (over 15-30 minutes), plus weekly trastuzumab 4 mg/kg IV (loading dose, over 90 minutes Day 1, Cycle 1 only) and 2 mg/kg IV (over 30-60 minutes on Days 1, 8, and 15) thereafter. Once 4 cycles of TC+H have been received, patients will continue with trastuzumab 6 mg/kg every 3 weeks to complete 1 year of anti-HER2 therapy as per the current standard of care. The anticipated time to study completion is 5 years.
  Other Names: trastuzumab

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) docetaxel/cyclophosphamide (brand names: Taxotere and Cytoxan, or TC) plus trastuzumab (brand name: Herceptin, or H) has HER2+ breast cancer.

ELIGIBILITY:
Inclusion Criteria:

A woman will be eligible for inclusion in this study if she meets all of the following criteria:

* Has HER2+ (IHC staining of 3+ [uniform, intense membrane staining of >30% of invasive tumor cells], or a FISH result of .6 HER2 gene copies per nucleus or a FISH ratio [HER2 gene signals to chromosome 17 signals] of >2.2; patients with equivocal FISH ratio results 1.8-2.2 are also eligible if 3+ IHC) (Appendix IX); Stage I, IIA, IIB, or IIIA T1-3N1-3M0 disease. At the discretion of the Treating Physician, patients with 4+ nodes with other factors such as patient choice, older age, preexisting cardiac disease with normal MUGA or ECHO may be enrolled into a separate subgroup.
* Has operable, histologically confirmed, invasive carcinoma of the breast.
* Has known ER and PR status
* Has adequate tumor specimen available for FISH analysis of TOP2A status (See Appendix VII)
* Has had no prior chemotherapy unless it was given >5 years ago for breast cancer or other cancer
* Has an ECOG Performance Status (PS) 0-1
* Age >18 to <70 years old.
* Has laboratory values of: See protocol for specific details
* Has aspartate aminotransferase (AST) or alanine aminotransferase (ALT) and alkaline phosphatase (ALP) within the ranges shown below. In determining eligibility the more abnormal of the 2 values (AST or ALT) should be used. See protocol for specific details
* Has complete surgical resection of the primary breast tumor: either lumpectomy or mastectomy with sentinel lymph node or axillary dissection.
* It has been <84 days since the date of definitive surgery, and there is adequate wound healing as determined by the Treating Physician
* Has no evidence of metastatic disease by physical examination and x-ray; appropriate scans as needed by each individual patient (eg, bone scan; abdominal, chest CT; PET or PET/CT; ultrasound; or MRI should indicate no evidence of metastatic disease.
* Has normal cardiac function as evidenced by a LVEF >50%, but must be within normal limits (WNL) by institutional standard, as determined by multiple gated acquisition (MUGA) scan. An echocardiogram (ECHO). The same modality must be used throughout the study to evaluate LVEF. Ejection fraction (EF) as determined by ECHO must be WNL by institutional standard.
* Has a negative serum pregnancy test within 7 calendar days prior to registration (female patients of childbearing potential [not surgically sterilized and between menarche and 1 year postmenopause]).
* If fertile, patient has agreed to use an acceptable method of birth control (barrier contraceptive) to avoid pregnancy for the duration of the study and for a period of 3 months thereafter
* Has signed a Patient Informed Consent Form
* Has signed a Patient Authorization Form

Exclusion Criteria:

A woman will be excluded from this study if she meets any of the following criteria:

* Has any evidence of disease following complete surgical resection of the primary tumor and metastatic workup
* Has Stage IIIB breast cancer (T4 disease; ie, patients with fixed tumors, peau d'orange skin changes, skin ulcerations, or inflammatory changes).
* Has Stage IV breast cancer (M1 disease on TNM staging system)
* Had prior chemotherapy for breast cancer or other cancer within the last 5 years (no neoadjuvant chemotherapy in this study is permitted)
* Has a history of severe hypersensitivity reaction to drugs formulated with polysorbate 80
* Has had a myocardial infarction (MI) within 6 months of trial enrollment, or has New York Heart Association (NYHA) Class II or greater heart failure (see Appendix III), uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic changes
* Has abnormal baseline MUGA (or ECHO) (<50%, or less than institutional LLN)
* Is receiving concurrent immunotherapy, hormonal therapy, or radiation therapy. Adjuvant hormonal therapy, if needed, may be given during radiation therapy and during treatment with trastuzumab after completion of chemotherapy.
* Is receiving concurrent investigational therapy or has received such therapy within the past 30 calendar days
* Has peripheral neuropathy >Grade 1
* Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious viral (including clinically defined AIDS), bacterial or fungal infection; or history of uncontrolled seizures, or diabetes, or CNS disorders deemed by the Treating Physician to be clinically significant, precluding informed consent
* Has active hepatitis B or hepatitis C with abnormal liver function tests (LFTs) or is known to be HIV positive
* Has a history of other malignancy within the last 5 years (except cured basal cell carcinoma of skin and carcinoma in situ of uterine cervix), which could affect the diagnosis or assessment of any of the study drugs
* Is an obese patient to whom the Treating Physician would not be comfortable administering full doses of study drugs as calculated by the BSA. Obese patients will be treated based on actual body weight. Obese patients treated with full doses based on actual BSA are eligible
* Is a pregnant or breastfeeding woman
* Is deemed unable to comply with requirements of study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2007-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Jones, MD, Principal Investigator — US Oncology Research
Locations (68):
- United States (68):
  - Birmingham Hematology and Oncology, Birmingham, Alabama
  - Hematology Oncology Associates, Phoenix, Arizona
  - Northern AZ Hematology & Oncology Associates, Sedona, Arizona
  - Arizona Oncology Associates DBA HOPE, Tucson, Arizona
  - Rocky Mountain Cancer Center-Rose, Denver, Colorado
  - Connecticut Oncology & Hematology, LLP, Torrington, Connecticut
  - Florida Cancer Institute, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Hematology Oncology Associates of IL, Chicago, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Hope Center, Terre Haute, Indiana
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Alliance Hematology Oncology P.A., Westminster, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Arch Medical Services, Inc., St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Hematology-Oncology Associates of NNJ, P.A., Morristown, New Jersey
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - Ruth Oratz MD, New York, New York
  - Interlakes Oncology Hematology, PC, Rochester, New York
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Texas Cancer Center-Abilene (South), Abilene, Texas
  - Texas Oncology, P.A.-Amarillo, Amarillo, Texas
  - Texas Cancer Center, Arlington, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology, P.A.-Bedford, Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Methodist Charlton Cancer Ctr., Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - El Paso Cancer Treatment Ctr, El Paso, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - Texas Oncology, P.A., Garland, Texas
  - Texas Oncology, P.A., Houston, Texas
  - Lake Vista Cancer Center, Lewisville, Texas
  - Longview Cancer Center, Longview, Texas
  - South Texas Cancer Center-McAllen, McAllen, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Allison Cancer Center, Midland, Texas
  - Texas Oncology-Odessa, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - San Antonio Tumor and Blood Clinic, San Antonio, Texas
  - HOAST-Medical Dr., San Antonio, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - Texas Oncology Cancer Center-Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology Cancer Care and Research, Waco, Texas
  - Texas Oncology PA, Webster, Texas
  - Texoma Cancer Center, Wichita Falls, Texas
  - Fairfax Northern VA Hem-Onc PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Onc and Hem Associates of SW VA, Inc., Salem, Virginia
  - Highline Medical Oncology, Burien, Washington
  - Puget Sound Cancer Center-Edmonds, Edmonds, Washington
  - Puget Sound Cancer Center-Seattle, Seattle, Washington
  - Cancer Care Northwest-South, Spokane, Washington
  - Northwest Cancer Specialists-Vancouver, Vancouver, Washington
  - Yakima Valley Mem Hosp/North Star Lodge, Yakima, Washington

REFERENCES:
- [Derived] Jones SE, Collea R, Paul D, Sedlacek S, Favret AM, Gore I Jr, Lindquist DL, Holmes FA, Allison MAK, Brooks BD, Portillo RM, Vukelja SJ, Steinberg MS, Stokoe C, Crockett MW, Wang Y, Asmar L, Robert NJ, O'Shaughnessy J. Adjuvant docetaxel and cyclophosphamide plus trastuzumab in patients with HER2-amplified early stage breast cancer: a single-group, open-label, phase 2 study. Lancet Oncol. 2013 Oct;14(11):1121-1128. doi: 10.1016/S1470-2045(13)70384-X. Epub 2013 Sep 3. PMID 24007746

RESULTS

PARTICIPANT FLOW:
Groups:
- TC+H: This is a nonrandomized, noncomparative, open-label Phase II study. On Day 1 of each 21-day cycle for a total of 4 cycles, patients will receive docetaxel (Taxotere) 75 mg/m^2 IV plus cyclophosphamide (Cytoxan) 600 mg/m^2 IV, plus weekly trastuzumab (Herceptin) 4 mg/kg IV (loading dose, Day 1, Cycle 1 only) and 2 mg/kg IV (on Days 1, 8, and 15) thereafter. Subsequent cycles of therapy will continue until a total of 4 cycles of TC+H have been completed. Then, patients will continue to receive trastuzumab 6 mg/kg every 3 weeks to complete 1 year of anti-HER2 therapy as per the current standard of care.
Period: Overall Study
Arm/Group | TC+H
Started | 493
Completed | 411
Not Completed | 82
Not completed — Adverse Event | 44
Not completed — Patient Request | 21
Not completed — Investigator Request | 2
Not completed — Disease Progression | 1
Not completed — Lost to Follow-up | 1
Not completed — Other | 13

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- TC+H: docetaxel (Taxotere), plus cyclophosphamide (Cytoxan), plus weekly trastuzumab (Herceptin)
Arm/Group | TC+H
Number analyzed (Participants) | 493
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 493
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 414
  Black | 36
  Hispanic | 27
  Asian | 12
  Indian | 1
  Other | 3
Region of Enrollment [Number; unit: participants]
  United States | 493

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS) Rate at 2 Years in TOP2A-amplified and in TOP2A-nonamplified HER2+ ESBC Patients Treated With TC+H.
Description: DFS was measured from the date of registration to either the date the patient was first recorded as having disease recurrence, or the date of death due to any causes before recurrence. If a patient had not recurred or died, DFS was censored at the date of last follow-up.
Time Frame: 2 years
Population: ITT population. Patients were excluded if their TOP2A amplification were unknown.
Measure: Number (95% Confidence Interval); unit: probability of disease-free survival
Groups:
- TOP2A-amplified Group: FISH ratio of TOP2A gene copy number was 2 or greater.
- TOP2A-nonamplified Group: FISH ratio of TOP2A gene copy number was less than 2.
Arm/Group | TOP2A-amplified Group | TOP2A-nonamplified Group
Number analyzed (Participants) | 190 | 248
probability of disease-free survival | 0.978 [0.942 to 0.992] | 0.979 [0.949 to 0.991]

2. Secondary Outcome: Overall Survival (OS) Rate at 2 Years in TOP2A-amplified and in TOP2A-nonamplified HER2+ ESBC Patients Treated With TC+H.
Description: OS is measured from the date of registration to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date.
Time Frame: 2 years
Population: ITT population. Patients were excluded if their TOP2A amplification were unknown.
Measure: Number (95% Confidence Interval); unit: probability of overall survival
Arm/Group | TOP2A-amplified Group | TOP2A-nonamplified Group
Number analyzed (Participants) | 190 | 248
probability of overall survival | 0.995 [0.962 to 0.999] | 0.988 [0.962 to 0.996]

3. Secondary Outcome: DFS by cMyc Expression in This Population of HER2+ ESBC Patients Treated With TC+H.
Description: as for outcome 1
Time Frame: 2 years
Population: ITT population. Patients were excluded if their cMYC amplification were unknown.
Measure: Number (95% Confidence Interval); unit: probability of disease-free survival
Groups:
- cMYC-amplified Group: FISH ratio of cMYC gene copy number was 2 or greater.
- cMYC-nonamplified Group: FISH ratio of cMYC gene copy number was less than 2.
Arm/Group | cMYC-amplified Group | cMYC-nonamplified Group
Number analyzed (Participants) | 99 | 337
probability of disease-free survival | 0.968 [0.904 to 0.990] | 0.981 [0.958 to 0.991]

4. Secondary Outcome: OS by cMyc Expression in This Population of HER2+ ESBC Patients Treated With TC+H.
Description: OS is measured from the date of randomization to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date.
Time Frame: 2 years
Population: ITT population. Patients were excluded if their cMYC amplification were unknown.
Measure: Number (95% Confidence Interval); unit: probability of overall survival
Arm/Group | cMYC-amplified Group | cMYC-nonamplified Group
Number analyzed (Participants) | 99 | 337
probability of overall survival | 0.990 [0.930 to 0.999] | 0.991 [0.972 to 0.997]

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Description: For treated patients only, assessed at each treatment visit.
Arm/Group | TC+H
Serious Adverse Events (participants affected / at risk) | 51/486
Other Adverse Events (participants affected / at risk) | 481/486
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TC+H (N=486)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BLOATING (Gastrointestinal disorders) | 1 (1)
BOWEL PERFORATION (Gastrointestinal disorders) | 1 (1)
CELLULITIS (Infections and infestations) | 4 (4)
CELLULITIS BREAST (Infections and infestations) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 5 (6)
DIARRHEA (Gastrointestinal disorders) | 5 (5)
DIVERTICULITIS (Infections and infestations) | 1 (1)
FEBRILE NEUTROPENIA (Infections and infestations) | 22 (23)
FEVER (General disorders) | 5 (5)
FIBRILLATION ATRIAL (Cardiac disorders) | 1 (1)
GASTRIC INFLAMMATION (Gastrointestinal disorders) | 1 (1)
HEPATIC ENZYMES INCREASED (Hepatobiliary disorders) | 1 (1)
HYPERSENSITIVITY REACTION (NOS) (Nervous system disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1)
INFECTION (Infections and infestations) | 1 (1)
LIVER FUNCTION TESTS MULTIPLE ABNORM (Hepatobiliary disorders) | 1 (1)
LUNG FIBROSIS INTERSTITIAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
MASTITIS (Infections and infestations) | 1 (1)
MUCOSITIS NOS (Infections and infestations) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (3)
NAUSEA AND VOMITING (Gastrointestinal disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (5)
PAIN (General disorders) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PULMONARY INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SHOCK (Nervous system disorders) | 1 (1)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (2)
THROMBOSIS ARTERIAL LEG (Vascular disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TC+H (N=486)
ALOPECIA (Skin and subcutaneous tissue disorders) | 339 (395)
ANEMIA (Blood and lymphatic system disorders) | 131 (227)
ANOREXIA (Gastrointestinal disorders) | 56 (69)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 66 (77)
CARDIAC INSUFFICIENCY (Cardiac disorders) | 29 (34)
CONSTIPATION (Gastrointestinal disorders) | 90 (112)
DIARRHEA (Gastrointestinal disorders) | 183 (276)
DYSGUESIA (Gastrointestinal disorders) | 73 (86)
EDEMA (Blood and lymphatic system disorders) | 86 (120)
FATIGUE (General disorders) | 284 (487)
FEVER (General disorders) | 42 (55)
GASTROESOPHAGEAL REFLUX (Gastrointestinal disorders) | 63 (68)
HEADACHE (General disorders) | 55 (67)
HOT FLASHES (General disorders) | 50 (59)
INSOMNIA (General disorders) | 49 (61)
LEUCOPENIA (Blood and lymphatic system disorders) | 84 (179)
MUCOSAL (Skin and subcutaneous tissue disorders) | 32 (39)
MUCOSITIS (Infections and infestations) | 89 (115)
MYALGIA (Musculoskeletal and connective tissue disorders) | 81 (96)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 34 (38)
NAUSEA (Gastrointestinal disorders) | 216 (315)
NEUROPATHY (Nervous system disorders) | 99 (125)
NEUTROPENIA (Blood and lymphatic system disorders) | 247 (597)
PAIN (General disorders) | 64 (91)
RASH (Skin and subcutaneous tissue disorders) | 104 (141)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 41 (46)
VOMITING (Gastrointestinal disorders) | 45 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No